CLINICAL TRIAL: NCT05001256
Title: Determination of Physical Activity Status and Adherence to the Mediterranean Diet in Adults and Related Health Outcomes
Status: Completed | Type: Observational
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Nezihe Otay Lule, Research assistant, University of Gaziantep
Other Study IDs: notaylule
Record Dates: First submitted 2021-08-05; First posted 2021-08-11 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Nutrition; Physical Activity; Chronic Disease; Obesity; Mediterranean Diet
Keywords: mediterranean diet; physical activity; obesity; chronic diseases
MeSH Terms: conditions — Motor Activity; Chronic Disease; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Individuals between the ages of 18-65 who applied to the physical therapy and rehabilitation outpatient clinic of a private hospital and voluntarily agreed to participate in the study will be included in the study. Written consent will be obtained from the participants.
  Participants' information will be recorded on a pre-prepared questionnaire containing structured questions. Questionnaire questioning will be applied to individuals through face-to-face interviews. The questionnaire form consists of three parts: 1. Sociodemographic characteristics, 2. Mediterranean Diet Adherence Scale (MEDAS), 3. International Physical Activity Questionnaire (IPAQ).
  Interventions: Other: questionnaire study

INTERVENTIONS:
Other: questionnaire study — Participants will be surveyed through face-to-face interviews.

SUMMARY:
A physically active life with adequate and balanced nutrition is essential for a healthy life. Unhealthy diet and being physically inactive are among the common risk factors that need to be corrected in order to maintain and improve health. The Mediterranean diet, first described by Angel Keys, is rich in plant foods such as grains, fruits, vegetables, legumes, oilseeds and olives; The main source of added oils is olive oil; moderate-high consumption of fish and seafood, moderate-level consumption of eggs, poultry and dairy products, and low-level red meat; It is a nutrition model with moderate intake of wine / fermented beverages (such as turnip, grape juice). Preferring vegetable oils instead of animal fats, preferring fish instead of red meat consumption, preferring low-fat / fat-free milk and dairy products, limiting the intake of simple sugar and refined carbohydrates, fruit rich in fiber and antioxidants in the Mediterranean diet, which is shown as an example of healthy nutrition today. It is thought that this type of nutrition can prevent the formation of chronic diseases due to features such as increasing vegetable consumption.

Determining the nutritional status and physical activity levels of individuals and their associated health outcomes; It is very important in terms of determining the current situation and determining the priority problems that need to be solved.

DETAILED DESCRIPTION:
A physically active life with adequate and balanced nutrition is essential for a healthy life. Unhealthy diet and being physically inactive are among the common risk factors that need to be corrected in order to maintain and improve health. In a cohort study of seven countries (USA, Finland, the Netherlands, Italy, the former Yugoslavia, Greece, and Japan) based on 25 years of follow-up and examining the relationship between dietary behaviors and mortality due to coronary heart disease, lower cardiovascular mortality rates were observed among participating countries in the Mediterranean region. . This has been attributed to traditional dietary behaviors such as high olive oil consumption in Greece, high fish consumption in Dalmatia (Croatia) and high vegetable consumption in Italy. Preferring vegetable oils instead of animal fats, preferring fish instead of red meat consumption, preferring low-fat/fat-free milk and dairy products, limiting simple sugar and refined carbohydrate intake, fruit rich in fiber and antioxidants in the Mediterranean diet, which is shown as an example of healthy nutrition today. It is thought that this type of nutrition can prevent the formation of chronic diseases due to the features such as increasing vegetable consumption. It is reported that low physical activity levels increase the risk of chronic diseases. Studies have shown that adherence to the Mediterranean diet is associated with lower BMI, total fat, and abdominal adiposity. It is also known that a decrease in body total fat rate is observed with physical activity. In addition, BMI values decrease with physical activity. With the changes in lifestyle habits in recent years, societies are moving away from the Mediterranean type of diet and becoming more and more sedentary. For this reason, it is very important to determine the current situation regarding the health outcomes related to the nutritional status and physical activity levels of the individuals, to determine the priority problems that need to be solved, and to raise the awareness of the society on this issue.

The aim of this study is to determine the adherence to the Mediterranean diet, physical activity status and related health outcomes of adult individuals who applied to the physical therapy outpatient clinic of a private hospital.

ELIGIBILITY:
Inclusion Criteria:

be between the ages of 18-65 having applied to the physical therapy outpatient clinic voluntarily agree to participate in research

Exclusion Criteria:

* be under the age of 18 be over 65

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals between the ages of 18-65 who applied to the physical therapy and rehabilitation outpatient clinic of a private hospital and voluntarily agreed to participate in the study will be included in the study.
Sampling Method: Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Mediterranean Diet Compliance Scale (MEDAS) | at baseline
  The 14-item Mediterranean Diet Adaptation Scale (MEDAS) will be used to determine the adaptation status of individuals to the Mediterranean diet. In the scale of adaptation to the Mediterranean diet, there are a total of 14 questions, 12 of which are about food consumption frequency and 2 are about food consumption habits. The score given for each question is 0 or 1 point. Then the scores are summed and the score is evaluated as ≤5 (low agreement), 6-9 (moderate agreement) and ≥10 (high agreement).
International Physical Activity Questionnaire (IPAQ) | at baseline
  The International Physical Activity Questionnaire (IPAQ) will be used to examine physical activity status. According to the IPAQ form, in which daily activities are evaluated as sitting, walking, moderate and vigorous activities and questioning the activity status in the past week, individuals are grouped as inactive (<600met), minimally active (600-3000met) and active (>3000met) according to their IPAQ scores.
obesity | at baseline
  Body mass index will be calculated by taking the person's height and body weight information.
  Waist and hip circumference measurements will also be made.
chronic disease | at baseline
  79 / 5000 Çeviri sonuçları Participants will be asked about the presence of a chronic disease diagnosed by the physician.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University, Şehitkamil, Gazi̇antep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No